CLINICAL TRIAL: NCT02759016
Title: A Phase Ib, Open Label, Single Arm, Multi-center, Dose Escalation Trial of Intravenous BI 836826 in Combination With Ibrutinib in Patients With Relapsed/Refractory Chronic Lymphocytic Leukemia
Brief Title: Intravenous BI 836826 in Combination With Ibrutinib in Relapsed/Refractory CLL Patients Who Have Been Pre-treated With at Least One Prior Line of Systemic Therapy, and Who Are Eligible for Treatment With Ibrutinib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1270.15
Record Dates: First submitted 2016-04-27; First posted 2016-05-03 (Estimated); Results first posted 2020-07-24 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Leukemia, Lymphocytic, Chronic, B-Cell
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — BI 836826; ibrutinib

ARMS (1):
- BI 836826 (Experimental): BI 836826 administered in combination with Standard of Care Ibrutinib
  Interventions: Drug: BI 836826; Drug: Ibrutinib

INTERVENTIONS:
Drug: BI 836826
Drug: Ibrutinib — Standard of Care

SUMMARY:
Intravenous BI 836826 in combination with ibrutinib in relapsed/refractory Chronic Lymphocytic Leukemia (CLL) patients who have been pre-treated with at least one prior line of systemic therapy, and who are eligible for treatment with ibrutinib. Objectives of the trial are to determine the recommended Phase 2 dose of BI 836826, and to document the safety and tolerability of BI 836826 when given in combination with ibrutinib

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of Chronic Lymphocytic Leukemia (CLL) established according to International Workshop Chronic Lymphocytic Leukemia (IWCLL) criteria.
* Relapsed or refractory CLL pre-treated with at least one prior line of systemic therapy for CLL.
* Indication for treatment consistent with IWCLL criteria, i.e. at least one of the following criteria should be met
* Evidence of progressive marrow failure as manifested by the development of, or worsening of, anemia and/or thrombocytopenia.
* Massive or progressive or symptomatic splenomegaly.
* Massive nodes or progressive or symptomatic lymphadenopathy.
* Progressive lymphocytosis in the absence of infection, with an increase in blood Absolute Lymphocyte Count (ALC) >=50% over a 2-month period, or a lymphocyte doubling time (LDT) of <6 months (as long as initial ALC was >=30000/µl).
* Autoimmune anemia and/or thrombocytopenia that is poorly responsive to corticosteroids or other standard therapy.
* Constitutional symptoms, defined as any one or more of the following disease-related symptoms or signs:
* unintentional weight loss of 10% or more within the previous 6 months
* significant fatigue
* fevers higher than 100.5°F or 38.0°C for >=2 weeks without other evidence of infection
* night sweats for > 1 month without evidence of infection
* Clinically quantifiable disease burden defined as at least one of the following:
* either ALC >10 000/µL, or
* measurable lymphadenopathy
* quantifiable bone marrow infiltration documented in a bone marrow biopsy during screening
* Resolution of all clinically relevant acute non-hematologic toxic effects of any prior antitumor therapy resolved to Grade <=1
* Baseline laboratory data as defined as:

Hemoglobin (Hb): >=8g/dL Absolute Neutrophil Count (ANC): >=1000/µL Platelet (PLT): >=25000/µL Glomerular Filtration Rate (GFR) or Creatinine Clearance: >=30ml/min Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT): <3 x Upper Limit of Normal (ULN) Bilirubin - total: <1.5 x ULN Activated Partial Thromboplastin Time (aPTT), Prothrombin Time (PT) or International Normalized Ratio (INR): <=1.5 x ULN PT <=1.5 x ULN, INR <=1.5

* Male or female patients. Women of childbearing potential must agree to use highly effective methods of birth control during the trial and for at least 1 year after the last dose of BI 836826 and 1 month after the last dose of ibrutinib.
* Eastern Cooperative Oncology Group (ECOG) performance score of 0 to 2.
* Age 18 years and older
* Eligible and able to secure sourcing for ibrutinib
* Written Informed Consent
* Further Inclusion criteria apply

Exclusion criteria:

* Known transformation of Chronic Lymphocytic Leukemia (CLL) to an aggressive B-cell malignancy at the time of screening
* Prior allogeneic stem cell transplant within one year or active graft vs. host disease.
* History of a non-CLL malignancy except for adequately treated in situ, stage 1 or 2 carcinoma in Complete Response (CR), or any other cancer that has been in CR for >=2 years after end of cancer treatment.
* Active, uncontrolled autoimmune cytopenia. Patients with autoimmune cytopenia which is controlled with corticosteroids at doses of <=20 mg prednisolone or equivalent may be enrolled.
* Previous CLL treatment with a CD37-targeting antibody or a CD37-antibody drug conjugate.
* Previous treatment with ibrutinib
* Previous treatment with another Bruton's Tyrosine Kinase (BTK) -inhibitor.
* Ongoing systemic immunosuppressive therapy other than corticosteroids.
* Active bacterial, viral, or fungal infection requiring systemic treatment at the time of study entry.
* Human Immunodeficiency Virus (HIV) infection
* Active hepatitis B or C as evidenced by detection of virus specific Deoxyribonucleic Acid (DNA) or Ribonucleic Acid (RNA).
* History of stroke or intracranial hemorrhage within 6 months prior to enrollment
* Chronic persistent atrial flutter or atrial fibrillation. Patients with intermittent atrial fibrillation may be enrolled if without episode for >= 6 months and without indication for anti-coagulation
* Requirement for chronic anticoagulation with warfarin or with direct oral anticoagulants at the time of screening.
* Chronic treatment (i.e. >7 days) with a strong Cytochrome P450 (CYP3A) inhibitor which cannot be terminated prior to the first dose of ibrutinib.
* Unstable angina pectoris, uncontrolled hypertension, uncontrolled asthma or other pulmonary disease
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial
* Further Exclusion criteria apply

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-06-23 (Actual); Primary Completion 2019-06-03 (Actual); Study Completion 2019-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (3):
- United States (3):
  - City of Hope, Duarte, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Oregon Health and Sciences University, Portland, Oregon

REFERENCES:
- See also: Related Info — https://trials.boehringer-ingelheim.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was planned to consist of 2 parts. First part was a Phase Ib, open-label, single arm, multi-center, dose escalation trial to determine the maximum tolerated dose and the recommended Phase II dose of intravenous BI 836826 in combination with ibrutinib. Original protocol planned a Phase II part which was not conducted.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that the subjects strictly met all inclusion and none of the exclusion criteria. Abbreviations: SD=Stable Disease, PR-MRDpos=Minimal Residual Disease positive Partial Response, PR-L=Partial Response with Lymphocytosis.
Groups:
- Dose Cohort BI 836826 100 Milligram (mg) + Ibrutinib; Dose Cohort BI 836826 200 Milligram (mg) + Ibrutinib: Participants underwent a 2-week run-in phase with ibrutinib prior to the start of BI 836826. In combination with ibrutinib (420 mg daily dose, orally administered) BI 836826 was administered intravenously as a rate controlled injection in 4-week cycles, every two weeks for the first 16 weeks (Cycles 1-4), and every 4 weeks starting at week 17 (Cycle 5) until week 48 (Cycle 12). BI 836826 was administered in Cycle 1 on day 1 (10 mg), days 2 and 8 (50% of the assigned dose on each day), day 15 (100% of the assigned dose), in Cycles 2-4 on days 1 and 15 of each cycle (100% of the assigned dose), in Cycles 5-12 on day 1 (100% of the assigned dose). Participants could have initiated 12 cycles with BI 836826 and could be treated with ibrutinib unless progression, unacceptable toxicity, or withdrawal of consent occurred earlier. Continued treatment beyond Cycle 12 (up to a maximum of 24 treatment cycles) was possible for participants with a pre-specified response status at end of Cycle 12.
Period: Overall Study
Arm/Group | Dose Cohort BI 836826 100 Milligram (mg) + Ibrutinib | Dose Cohort BI 836826 200 Milligram (mg) + Ibrutinib
Started (Assigned to combination treatment BI 836826 and ibrutinib) | 4 | 3
Treated With BI 836826 and Ibrutinib | 3 | 3
Completed | 0 | 0
Not Completed | 4 | 3
Not completed — Not treated with BI 836826 | 1 | 0
Not completed — Progressive disease | 1 | 0
Not completed — SD, PR-MRDpos or PR-L | 0 | 2
Not completed — Other not defined above | 2 | 1

BASELINE CHARACTERISTICS:
Population: The Treated Set (TS) included all participants who initiated at least one administration of BI 836826. The TS was used for all planned safety and efficacy analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Cohort BI 836826 100 Milligram (mg) + Ibrutinib | Dose Cohort BI 836826 200 Milligram (mg) + Ibrutinib | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.0 (4.4) | 66.0 (8.5) | 69.5 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase 2 Dose of BI 836826 in Combination With Ibrutinib
Description: The Recommended Phase 2 Dose (RP2D ) of BI 836826 in combination with ibrutinib would be either the Maximum Tolerated Dose (MTD) or a lower dose and would be determined by the safety review committee based on safety and efficacy considerations.
Time Frame: First treatment cycle, 4 weeks from first administration of BI 836826.
Population: As the study was prematurely discontinued, recruitment of participants into the dose escalation part was not fully completed, the MTD was not reached and hence the RP2D could not be determined.
Groups:
- BI 836826 + Ibrutinib: Treatment group "BI 836826 + ibrutinib" comprises all dose cohorts during the dose escalation phase, that is, "Dose cohort BI 836826 100 mg + ibrutinib" and "Dose cohort BI 836826 200 mg + ibrutinib".
  Participants underwent a 2-week run-in phase with ibrutinib prior to the start of BI 836826. In combination with ibrutinib (420 mg daily dose, orally administered) BI 836826 was administered intravenously in Cycle (=4 weeks) 1 on day 1 (10 mg), days 2 and 8 (50% of the assigned dose on each day), day 15 (100% of the assigned dose), in Cycles 2-4 on days 1 and 15 of each cycle (100% of the assigned dose), in Cycles 5-12 on day 1 (100% of the assigned dose). Participants could have initiated 12 cycles with BI 836826 and could be treated with ibrutinib unless progression, unacceptable toxicity, or withdrawal of consent occurred earlier. Continued treatment beyond Cycle 12 (up to 24 treatment cycles) was possible for participants with a pre-specified response status at end of Cycle 12.
Arm/Group | BI 836826 + Ibrutinib
Number analyzed (Participants) | 0

2. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) During the First Treatment Cycle
Description: Number of participants with Dose Limiting Toxicities (DLTs) during the first treatment cycle. DLT was defined as any non-hematologic adverse event (AE) of Grade ≥ 3 related to BI 836826 and/or ibrutinib except infusion-related reaction (any Grade), Grade 3 Aspartate Aminotransferase (AST)- and/or Alanine Aminotransferase (ALT) elevation without concomitant bilirubin, elevation or any other asymptomatic Grade 3 laboratory abnormality with spontaneous recovery within 1 week. The following hematologic AEs related to BI 836826 and/or ibrutinib were considered DLT: Grade 4 neutropenia with concomitant infection, Grade 4 febrile neutropenia, and Grade 3 febrile neutropenia not resolving within 72 hours with appropriate treatment (antibiotics, antivirals, antifungals, growth factor support), Grade 4 thrombocytopenia with clinically significant bleeding, Grade 4 anemia, any Grade 5 hematologic AE.
Time Frame: First treatment cycle, 4 weeks from first administration of BI 836826.
Population: All participants who were documented to have initiated at least one dose of BI 836826 and were not replaced for the Maximum Tolerated Dose (MTD) evaluation.
Measure: Number; unit: Participants
Arm/Group | Dose Cohort BI 836826 100 Milligram (mg) + Ibrutinib | Dose Cohort BI 836826 200 Milligram (mg) + Ibrutinib
Number analyzed (Participants) | 3 | 3
Participants | 0 | 0

3. Secondary Outcome: Maximum Tolerated Dose of BI 836826 in Combination With Ibrutinib
Description: To determine the Maximum Tolerated Dose (MTD) of BI 836826 in combination with ibrutinib, participants were entered sequentially into dose cohorts starting at 100 mg of BI 836826 and escalating to the MTD in combination with ibrutinib (fixed dose of 420 mg daily). Stepwise dose escalation of BI 836826 was guided by a Bayesian Logistic Regression Model (BLRM) with overdose control. The BLRM estimates the MTD by updating estimates of the probability of observing a Dose Limiting Toxicity (DLT) in the first treatment cycle (4 weeks) for each dose level as participant information becomes available. The MTD would be considered reached if the following criteria were fulfilled. The posterior probability of the true DLT rate in the target interval [0.16 - 0.33) of the MTD is above 0.50 or at least 15 participants have been treated in the study, of which at least 6 at the MTD.
Time Frame: First treatment cycle, 4 weeks from first administration of BI 836826.
Population: As the study was prematurely discontinued, recruitment of participants into the dose escalation part was not fully completed and the MTD was not reached.
Arm/Group | BI 836826 + Ibrutinib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: On-treatment period + Residual Effect Period, that is, from first administration of BI 836826 until the end of the Residual Effect Period (30 days after the last infusion of BI 836826), up to 22 treatment cycles = 22 * 4 weeks + 30 days = 646 days.
Description: All participants who initiated at least one administration of BI 836826.
Arm/Group | Dose Cohort BI 836826 100 Milligram (mg) + Ibrutinib | Dose Cohort BI 836826 200 Milligram (mg) + Ibrutinib
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 2/3 | 3/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Cohort BI 836826 100 Milligram (mg) + Ibrutinib (N=3) | Dose Cohort BI 836826 200 Milligram (mg) + Ibrutinib (N=3)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Pseudomonal bacteraemia (Infections and infestations) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Cohort BI 836826 100 Milligram (mg) + Ibrutinib (N=3) | Dose Cohort BI 836826 200 Milligram (mg) + Ibrutinib (N=3)
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Lip swelling (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Oral pain (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 2
Malaise (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 0
Bronchitis (Infections and infestations) | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 1
Nail infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 3
Urinary tract infection (Infections and infestations) | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Incision site pain (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 1
Blood creatinine increased (Investigations) | 2 | 0
White blood cell count decreased (Investigations) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Development of BI 836826 was discontinued (strategic decision). Recruitment was subsequently terminated, the Phase II part of the trial was eliminated from the protocol, participants on treatment were allowed to complete the trial as per protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-07-30): https://cdn.clinicaltrials.gov/large-docs/16/NCT02759016/SAP_001.pdf
  • Study Protocol (2018-07-18): https://cdn.clinicaltrials.gov/large-docs/16/NCT02759016/Prot_002.pdf